CLINICAL TRIAL: NCT04999657
Title: A Prospective, Multi-center, Randomized Controlled, Double-blind, Superiority Clinical Trial Evaluating the Safety and Efficacy of a Non-invasive Low-frequency Tibial Nerve Stimulator for the Treatment of Overactive Bladder
Brief Title: Evaluation of the The Neuromodulation System for the Treatment of Overactive Bladder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtecx Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMK03025P
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Device: Non-invasive low-frequency tibial nerve stimulator
  Interventions: Device: Non-invasive low-frequency tibial nerve stimulator (TNS-01)
- Sham (Sham Comparator): Device: Non-invasive low-frequency tibial nerve stimulator (same device operation without real current output)
  Interventions: Device: Non-invasive low-frequency tibial nerve stimulator (TNS-01)

INTERVENTIONS:
Device: Non-invasive low-frequency tibial nerve stimulator (TNS-01) — The investigational device is a transcutaneous electrical nerve stimulation (TENS) device that is designed to provide stimulation to the nerves at the site of application via surface electrodes temporarily adhered to the skin.

SUMMARY:
To evaluate the efficacy and safety of non-invasive tibial nerve stimulator for the treatment of overactive bladder under the premise of ensuring the safety of the subjects and ensuring the scientific nature of the clinical trial. The primary safety endpoint will be device-related adverse events. The primary effectiveness endpoint will be the improvement value of overactive bladder symptom score (OABSS) after 12-week treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged between 18 and 80 years old (including 18 and 80 years old)；
2. Individual with primary OAB, or with OAB symptoms, satisfies one of the following conditions:

   ① Urinary urgency: sudden and strong desire to urinate, and it is difficult to be subjectively suppressed and delayed urination ;

   ② Urge urinary incontinence: accompanied with urinary urgency or immediately after urinary urgency ;

   ③ Urination frequency: adults urination frequency ≥8 times during the daytime，≥2 times at night, and each urine volume <200 ml .
3. Individual meets the diagnostic criteria of OAB: According to the OABSS questionnaire, urgency score ≥2 points, total score ≥3 points, and symptoms duration ≥3 months;
4. Individual newly diagnosed with OAB have not been medicated, or is able to stop taking OAB-related drugs (M receptor block, β3 receptor agonists) for at least 2 weeks prior to enrollment;
5. The subject has autonomy and can go to the toilet independently;
6. Individual is ambulatory and able to use the toilet independently;
7. Individual is capable and willing to participate in the study and provide the written informed consent.

Exclusion Criteria:

1. Woman is pregnant or lactating, or woman of childbearing age who plans to become pregnant during the study period;
2. Individual has Stress Urinary Incontinence (SUI);
3. Individual has obvious urinary obstruction due to various reasons accompanied by residual urine volume> 100 ml;
4. Individual has an implanted pacemaker, embedded cardioverter defibrillator, or other electrical medical devices (including sacral neuromodulation (SNM) devices)
5. Individual has uncured urinary system infection;
6. Individual has urinary calculus resulting in lower urinary tract symptoms;
7. Individual has congenital urinary tract malformations causing uncured lower urinary tract symptoms;
8. Individual has uncured cancers;
9. Individual had undergone lower urinary tract surgery within 3 months;
10. Individual has neurological diseases or injuries accompanied with uncured lower urinary tract symptoms;
11. Individual has skin breakage, malignant tumor or acute purulent inflammation on the surface of the plantar where the electrode pads are to be placed;
12. Individual has participated in other drug clinical trials medical dev within 3 months, or participated in other ice clinical trials within 30 days;
13. Individual is deemed unsuitable for enrollment in the study by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
The change of overactive bladder symptom score (OABSS) after 12-week treatment compared with baseline | 12 weeks
  OABSS is evaluated via 3-day voiding diary and urinary voiding events of the previous week at week 0, 4, 8 and 12 after treatment. Evaluate OABSS improvement from baseline after 12 weeks of treatment and compared between the Treatment and the Control groups

CONTACTS AND LOCATIONS:
Overall Officials: Yaoguang Zhang, MD, Principal Investigator — Beijing Hospital
Locations (7):
- China (7):
  - Beijing Hospital, Beijing, Beijing Municipality
  - West China Hospital, Chengdu
  - Nan Fang Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Shanghai Fifth People's Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - The First Affiliated Hospital of XI'AN JiaoTong University, Xi'an

REFERENCES:
- [Derived] Zhang Z, Liu M, Wang Y, Wu P, Zhu Y, Han B, Xu Z, Li X, Shi C, Zhang J, Luo D, Shi G, Zhang Y. Efficacy and safety of non-invasive low-frequency tibial nerve stimulator in overactive bladder. Eur J Med Res. 2025 Jan 20;30(1):40. doi: 10.1186/s40001-024-02262-z. PMID 39833952